CLINICAL TRIAL: NCT05101109
Title: A Phase 1 Dose Escalation and Expansion Study of ABL501, a Bispecific Antibody of PD-L1 and LAG-3 as a Single Agent in Subjects With Any Progressive, Locally Advanced (Unresectable) or Metastatic Solid Tumors
Brief Title: Study to Evaluate the Safety and Tolerability of ABL501, and to Determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of ABL501 in Subjects With Any Progressive, Locally Advanced (Unresectable) or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ABL Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABL501-1001
Record Dates: First submitted 2021-10-06; First posted 2021-11-01 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumor
Keywords: LAG-3; PD-L1; Immune oncology; solid tumor; bispecific antibody
MeSH Terms: interventions — Antibodies, Bispecific

STUDY DESIGN:
Intervention Model Description: Drug: ABL501
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABL501 (Experimental): ABL501 will be administered biweekly of every 28-day cycle in the dose-escalation.
  Interventions: Drug: ABL501

INTERVENTIONS:
Drug: ABL501 — ABL501 will be administered biweekly of every 28-day cycle in the dose-escalation. The dosing interval to be used in the dose-expansion part will be re-evaluated based on the emerging safety and PK data from the dose-escalation part of the study.
  Other Names: Bispecific antibody for LAG-3 and PD-L1

SUMMARY:
This is a first-in-human (FIH) phase 1 open-label, multicenter, multiple-dose, dose-escalation and dose-expansion study of ABL501 to evaluate the safety, tolerability, MTD and/or RP2D, PK, immunogenicity, preliminary anti-tumor activity, and the PD effect of ABL501 in subjects with any progressive locally advanced (unresectable) or metastatic solid tumors. This study included 2 parts; a dose-escalation part and a dose expansion part.

DETAILED DESCRIPTION:
This is consisted with dose-escalation and dose-expansion study of ABL501 to evaluate the safety, tolerability, MTD and/or RP2D, PK, immunogenicity, anti-tumor activity, and the PD effect of ABL501 in subjects with any progressive locally advanced (unresectable) or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed any progressive, locally advanced (unresectable), or metastatic solid tumors that have relapsed or are refractory following the last line of treatment and for which prior standard therapy has been ineffective, standard therapy does not exist, or is not considered appropriate.
* Subjects with adverse events(AEs) excluding alopecia or Grade 2 toxicities that are deemed stable or irreversible (e.g., peripheral neuropathy) from prior therapy that have improved to Grade 1 or the baseline grade more than 14 days prior to the first administration of study drug.
* Subject with adequate hematologic, hepatic, and renal functions confirmed based on the screening laboratory test within 7 days prior to the first administration of ABL501

Exclusion Criteria:

* Subjects has received prior anticancer monoclonal antibody treatment or investigational therapy within 28 days prior to the first administration of ABL501 or who has recovered (i.e., =<Grade 1 or at baseline grade) from AEs due to previously administered agent more than 14 days prior to ABL501 administration.
* Subject has had prior chemotherapy or radiation therapy within 2 weeks or targeted small molecule therapy within 5 half-lives prior to the first administration of study drug or has not recovered (i.e., =<Grade 1 or at baseline grade) from AEs due to previously administered agent more than 14 days prior to ABL501 administration
* Subject discontinued from prior immunomodulatory therapy due to any intolerable immune-related AE(s) (irAEs) requiring systemic steroid treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Number of subjects with dose-limiting toxicities (DLT) | from Day 1 until Day 28
  Number of subject with dose-limiting toxicities (DLT)
Number of subjects who experience with TEAEs, SAEs, irAEs and IRRs | From Day 1 until confirmed CR, disease progression, unacceptable toxicity or subject/investigator's decision to terminate the study participation, assessed up to 24 months
  Number of subjects who experience with Treatment-emergent adverse events (TEAEs), Serious adverse events (SAEs), immune-related adverse events (irAEs) and infusion related reactions (IRRs)
Number of subjects who experience with treatment-related TEAEs, SAEs, irAEs and IRRs | From Day 1 until confirmed CR, disease progression, unacceptable toxicity or subject/investigator's decision to terminate the study participation, assessed up to 24 months
  Number of subjects who experience with treatment-related Treatment-emergent adverse events (TEAEs), Serious adverse events (SAEs), immune-related adverse events (irAEs) and infusion related reactions (IRRs)
Number of subjects who experience with clinically significant changes in laboratory values | From Day 1 until confirmed CR, disease progression, unacceptable toxicity or subject/investigator's decision to terminate the study participation, assessed up to 24 months
  Number of subjects who experience with clinically significant changes in laboratory values

SECONDARY OUTCOMES:
Pharmacokinetic profile of ABL501 | From Day 1 until confirmed CR, disease progression, unacceptable toxicity or subject/investigator's decision to terminate the study participation, assessed up to 24 months
  serum concentration of ABL501 will be collected and analyzed to evaluate the PK of ABL501
Objective Response Rate (ORR) | From Day 1 until confirmed CR, disease progression, unacceptable toxicity or subject/investigator's decision to terminate the study participation, assessed up to 24 months
  Proportion of subjects with best overall response of complete response (CR) or partial response (PR) per RECIST v1.1
number of subject with anti-drug antibodies (ADAs) | From Day 1 until confirmed CR, disease progression, unacceptable toxicity or subject/investigator's decision to terminate the study participation, assessed up to 24 months
  Incidence of anti-drug antibodies (ADAs) will be analyzed to evaluate the immunogenicity of ABL501

CONTACTS AND LOCATIONS:
Overall Officials: Sangmi Lee, Study Director — Clinical development team
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sung E, Ko M, Won JY, Jo Y, Park E, Kim H, Choi E, Jung UJ, Jeon J, Kim Y, Ahn H, Choi DS, Choi S, Hong Y, Park H, Lee H, Son YG, Park K, Won J, Oh SJ, Lee S, Kim KP, Yoo C, Song HK, Jin HS, Jung J, Park Y. LAG-3xPD-L1 bispecific antibody potentiates antitumor responses of T cells through dendritic cell activation. Mol Ther. 2022 Aug 3;30(8):2800-2816. doi: 10.1016/j.ymthe.2022.05.003. Epub 2022 May 6. PMID 35526096